CLINICAL TRIAL: NCT03988400
Title: Development of Sensory Augmentation Methods to Improve Post-stroke Gait Stability
Brief Title: Sensory Augmentation Methods in Stroke
Acronym: SAM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3146-R
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: stroke; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an Experimental (n=22) or Control (n=22) group. These groups will differ only in terms of how vibration is delivered to the hip musculature during training sessions. In the Experimental group, vibration magnitude will be controlled by the real-time mechanical state of the user's body. In the Control group, vibration magnitude will be randomly varied.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensory augmentation (Experimental): Participants will complete 8 training sessions over 4 weeks, in which they walk on a treadmill at their self-selected speed. During training sessions, the magnitude of the vibration delivered over the hip abductor musculature will scale with the mechanical state of the pelvis at the start of each step. For example, if the step begins with the pelvis far mediolaterally from the stance foot, the swing leg hip abductors will receive strong vibration. If instead the step begins with the pelvis close mediolaterally to the stance foot, the stance hip abductors will receive strong vibration.
  Interventions: Behavioral: Sensory Augmentation
- Random vibration (Active Comparator): Participants will complete 8 training sessions over 4 weeks, in which they walk on a treadmill at their self-selected speed. During training sessions, the magnitude of the vibration applied to the hip abductors will vary randomly (following a normal distribution) on a step-by-step basis.
  Interventions: Behavioral: Random Vibration

INTERVENTIONS:
Behavioral: Sensory Augmentation — Participants will complete 8 training sessions over 4 weeks, in which they walk on a treadmill at their self-selected speed. During training sessions, the magnitude of the vibration delivered over the hip abductor musculature will scale with the mechanical state of the pelvis at the start of each step. For example, if the step begins with the pelvis far mediolaterally from the stance foot, the swing leg hip abductors will receive strong vibration. If instead the step begins with the pelvis close mediolaterally to the stance foot, the stance hip abductors will receive strong vibration.
  Arms: Sensory augmentation
Behavioral: Random Vibration — Participants will complete 8 training sessions over 4 weeks, in which they walk on a treadmill at their self-selected speed. During training sessions, the magnitude of the vibration applied to the hip abductors will vary randomly (following a normal distribution) on a step-by-step basis.
  Arms: Random vibration

SUMMARY:
Many chronic stroke survivors have poor walking balance, contributing to an increased risk of falls and fear of falling. One factor contributing to these balance deficits is a reduced ability to place the feet appropriately when walking. This study investigates whether enhancing the sensory information available to chronic stroke survivors while they walk improves their foot placement accuracy and balance.

DETAILED DESCRIPTION:
The objective of this project is to test a method of providing real-time augmentation of hip proprioceptive feedback during post-stroke walking. The sensory information available to participants will be augmented by providing vibration of the hip abductor musculature that is scaled to the near-real-time mechanical state of their body. The central hypothesis is that augmented proprioception will improve participants' perception of their body's motion, thus increasing the mechanics-dependent modulation of foot placement, an important gait stabilization strategy. This clinical trial will establish the safety, feasibility, and efficacy of a rehabilitation intervention centered on repeated exposure to sensory augmentation during gait. Specifically, participants in the experimental group will complete training sessions twice a week for four weeks in which they receive sensory augmentation during ~30 minutes of treadmill walking. Participants in the activity-matched control group will perform the same task, except the hip vibration will be randomly delivered, not linked to the body's actual mechanical state. Changes in walking balance and foot placement accuracy will be quantified over the course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Experience of a stroke 6 months prior to participation
* Gait speed of at least 0.2 m/s
* Ability to walk on a treadmill without a cane or walker
* Provision of informed consent

Exclusion Criteria:

* Evidence of cerebellar damage
* Resting blood pressure higher than 220/110 mm Hg
* History of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living
* Preexisting neurological disorders or dementia
* Legal blindness or severe visual impairment
* History of DVT or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Orthopedic injuries or conditions (e.g. joint replacements) in the lower extremities with the potential to alter the gait pattern

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C. Dean, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the assessment sessions (Week 0 and Week 4) will be shared. Specifically, this will include gait biomechanics data (e.g. the partial correlation between mediolateral foot placement and mediolateral pelvis displacement), Functional Gait Assessment scores, Activity-specific Balance Confidence scores, overground gait speeds, and self-reported fear of falling.
Supporting Information: Study Protocol
Time Frame: Data will be shared 1-month following publication of summary data, and will be shared in perpetuity.
Access Criteria: No criteria are anticipated to restrict who de-identified data will be shared with.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled into this study between April of 2022 and March of 2023. All participants were recruited from the RESTORE database at the Medical University of South Carolina.
Pre-assignment Details: Participants completed an initial assessment session prior to their assignment to a study arm/group. No qualified participants were enrolled into the study, but then excluded from the study before group assignment.
Period: Overall Study
Arm/Group | Sensory Augmentation | Random Vibration
Started | 22 | 22
Completed | 20 | 21
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Macular degeneration, unrelated to study procedures. | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Information is presented for all participants who enrolled in this intervention study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensory Augmentation | Random Vibration | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 57 (12) | 60 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mechanics-dependent Adjustment of Paretic Foot Placement [Mean (Standard Deviation); unit: Unitless (correlation coefficient)] — This measure is calculated as the partial correlation between mediolateral pelvis displacement at the start of a paretic step and mediolateral foot placement at the end of the paretic step, accounting for mediolateral velocity of the pelvis. This biomechanical measure of an important gait balance strategy is calculated using data collected from motion capture during treadmill walking.
  Unitless (correlation coefficient) | -.145 (.253) | -.043 (.236) | -.094 (.247)
Mechanics-dependent adjustment of Non-paretic Foot Placement [Mean (Standard Deviation); unit: Unitless (correlation coefficient)] — This measure is calculated as the partial correlation between mediolateral pelvis displacement at the start of a non-paretic step and mediolateral foot placement at the end of the non-paretic step, accounting for mediolateral velocity of the pelvis. This biomechanical measure of an important gait balance strategy is calculated using data collected from motion capture during treadmill walking.
  Unitless (correlation coefficient) | -.192 (.231) | -.075 (.254) | -.134 (.247)
Fear of Falling [Count of Participants; unit: Participants] | 8 | 11 | 19
Functional Gait Assessment score [Mean (Standard Deviation); unit: units on a scale] — The minimum value is 0, the maximum value is 30, and higher scores indicate a better outcome.
  units on a scale | 15.27 (5.81) | 15.23 (4.66) | 15.25 (5.20)
Activities-specific Balance Confidence scale score [Mean (Standard Deviation); unit: units on a scale] — The minimum value is 0, the maximum value is 100, and higher scores indicate a better outcome.
  units on a scale | 65.0 (20.0) | 64.2 (19.7) | 64.6 (19.6)
Self-selected overground walking speed [Mean (Standard Deviation); unit: meter per second] | 0.82 (0.30) | 0.75 (0.27) | 0.79 (0.29)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Related or Serious Adverse Events
Description: The investigators will monitor the safety of the intervention by quantifying the percentage of participants who experience an adverse event potentially related to the intervention (e.g. skin irritation; falls) or any serious adverse event (e.g. hospitalization; death). This information is gathered through participant self-report, or through communication with participant caregiver if necessary.
Time Frame: Cumulative over the course of the 4-week intervention
Population: Analysis was performed on all participants who began the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 22 | 22
Participants | 1 | 0
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 1, Fisher Exact — The a priori threshold for statistical significance was 0.05

2. Primary Outcome: Number of Training Sessions Attended
Description: The investigators will assess participant adherence as the number of training sessions attended (out of a maximum possible number of 8).
Time Frame: Cumulative over the course of the 4-week intervention
Population: Data was analyzed for all participants who completed the final assessment session.
Measure: Median (Full Range); unit: Visits attended
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
Visits attended | 7 [3 to 8] | 8 [6 to 8]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.017, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05

3. Primary Outcome: Intervention Feasibility (Drop-out)
Description: The investigators will assess participant drop-out as the number of participants who do not attend the final Assessment Session.
Time Frame: 4-weeks
Population: Data from all participants enrolled in this study was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 22 | 22
Participants | 2 | 1
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 1, Fisher Exact — The a priori threshold for statistical significance was 0.05

4. Primary Outcome: Change in Mechanics-dependent Adjustment of Paretic Foot Placement
Description: The primary effectiveness measure will be the change in participants' gait stabilization strategy over the course of the 4-week intervention. This will be quantified as the partial correlation between paretic mediolateral foot placement and mediolateral pelvis displacement at the start of the step over a 2-minute period of walking. The investigators will calculate the change in this metric from the initial (Week 0) assessment session to the final (Week 4) assessment session.
Time Frame: 4-weeks
Population: Analyses included participants who completed the final assessment session.
Measure: Mean (95% Confidence Interval); unit: Unitless (correlation coefficient)
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
Unitless (correlation coefficient) | 0.078 [0.002 to 0.154] | 0.054 [-0.053 to 0.160]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.72, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

5. Secondary Outcome: Intervention Feasibility (Walking Time)
Description: The investigators will quantify the total walking time across all training sessions (out of a maximum possible 312 minutes).
Time Frame: Cumulative over the course of the 4-week intervention
Population: Data was analyzed for all participants who completed the final assessment session.
Measure: Median (Full Range); unit: Minutes of walking
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
Minutes of walking | 144 [72 to 297] | 255 [75 to 312]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.001, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

6. Secondary Outcome: Change in Fear of Falling
Description: The investigators will assess the change in fear of falling (identified using a yes/no question of "do you have a fear of falling?") from the initial (Week 0) assessment session to the final (Week 4) assessment session.
Time Frame: 4-weeks
Population: Analysis was performed for all participants who completed the final assessment session.
Measure: Count of Participants; unit: Participants
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
Participants
  Fear of falling in initial assessment session | 8 | 10
  Fear of falling in final assessment session | 8 | 9
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05

7. Secondary Outcome: Change in Functional Gait Assessment Score
Description: The investigators will quantify the change in Functional Gait Assessment score from the initial (Week 0) assessment session to the final (Week 4) assessment session. The initial score will be subtracted from the final score. The minimum value is 0, the maximum value is 30, and higher scores indicate a better outcome.
Time Frame: 4-weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
score on a scale | 0.8 [-0.5 to 2.0] | 1.7 [0.7 to 2.7]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.25, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

8. Secondary Outcome: Change in Activity-specific Balance Confidence Score
Description: The investigators will quantify the change in Activity-specific Balance Confidence score from the initial (Week 0) assessment session to the final (Week 4) assessment session. The initial score will be subtracted from the final score. The minimum value is 0, the maximum value is 100, and higher scores indicate a better outcome.
Time Frame: 4-weeks
Population: Data was analyzed for participants who completed the final assessment session.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
score on a scale | 1.0 [-3.2 to 5.1] | 2.1 [-1.8 to 6.0]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.69, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

9. Secondary Outcome: Change in Overground Self-selected Gait Speed
Description: The investigators will quantify the change in overground self-selected gait speed from the initial (Week 0) assessment session to the final (Week 4) assessment session. The initial score will be subtracted from the final score.
Time Frame: 4-weeks
Population: Data was analyzed for participants who completed the final assessment session.
Measure: Mean (95% Confidence Interval); unit: meters per second
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
meters per second | 0.01 [-0.04 to 0.05] | 0.05 [0.00 to 0.10]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.20, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

10. Post Hoc Outcome: Change in Mechanics-dependent Adjustment of Non-paretic Foot Placement
Description: This not pre-planned effectiveness measure is the change in participant's gait stabilization over the course of the 4-week intervention for steps taken with the non-paretic leg. This was quantified as the partial correlation between non-paretic mediolateral foot placement and mediolateral pelvis displacement at the start of the step over a 2-minute period of walking. The change in this metric was calculated from the initial (Week 0) assessment session to the final (Week 4) assessment session. The initial score was subtracted from the final score.
Time Frame: 4-weeks
Population: Analyses included participants who completed the final assessment session.
Measure: Mean (95% Confidence Interval); unit: Unitless (correlation coefficient)
Arm/Group | Sensory Augmentation | Random Vibration
Number analyzed (Participants) | 20 | 21
Unitless (correlation coefficient) | 0.073 [-0.020 to 0.167] | 0.037 [-0.067 to 0.141]
Statistical Analysis 1: Comparison: Sensory Augmentation vs Random Vibration; Test type: Superiority; p = 0.62, t-test, 2 sided — The a priori threshold for statistical significance was 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the period spanning from the participant's initial assessment session through their final assessment session. This duration was approximately 5 weeks (initial assessment session; 4 weeks of training; final assessment session).
Description: The investigators followed the Clinicaltrials.gov definition.
Arm/Group | Sensory Augmentation | Random Vibration
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensory Augmentation (N=22) | Random Vibration (N=22)
Stroke (Vascular disorders) | 1 (1) | 0 (0) — One participant experienced a stroke while enrolled in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03988400/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03988400/ICF_000.pdf